CLINICAL TRIAL: NCT05193981
Title: Role of Homocysteine Metabolism, Endothelial Function and Microvascular Rarefaction on Renal Disease Severity and Progression in ADPKD
Brief Title: A Study to Evaluate Homocysteine Metabolism and Endothelial Function in ADPKD
Acronym: HCY
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Maria V. Irazabal Mira, Principal Investigator, Mayo Clinic
Other Study IDs: 20-005312; 1R01DK128017-01 (NIH)
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Autosomal Dominant Polycystic Kidney Disease (ADPKD); Endothelial function; Endothelial dysfunction; Homocysteine metabolism; Oxidative stress; NADPH oxidase 4 (NOX4)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a previous diagnosis of ADPKD: Patients that have been diagnosed with ADPKD and meet the study's inclusion criteria

SUMMARY:
The purpose of this study is to assess homocysteine metabolism and systemic endothelial function at the early stages of the disease and determine the prognostic value of homocysteine, related metabolites, and markers of endothelial function and injury to estimate renal disease severity and progression in patients with early Autosomal Dominant Polycystic Kidney Disease (ADPKD).

DETAILED DESCRIPTION:
ADPKD is a devastating systemic disorder characterized by progressive development and enlargement of bilateral renal cysts, often leading to renal failure. Disease severity and progression vary widely among patients. Large phenotypic variability, incomplete understanding of underlying mechanisms, and lack of suitable biomarkers challenge potential therapies' identification, implementation, and evaluation.

In ADPKD, systemic endothelial dysfunction (ED), characterized by an imbalance between vasodilating (particularly nitric oxide, NO) and vasoconstricting substances, develops early and correlates with renal disease severity. It has been previously associated with decreased NO availability, but NO abnormalities' mechanisms are still poorly understood. Endothelium-dependent, NO-mediated vasodilation is impaired in subjects with hyperhomocysteinemia, suggesting that NO availability is decreased in these subjects. Increased plasma levels of homocysteine have been reported in patients with ADPKD and preserved kidney function, likely contributing to a reduction in NO bioavailability. The mechanisms underlying increased homocysteine in ADPKD are not known. Furthermore, whether systemic endothelial function and injury or homocysteine levels can predict renal disease severity and progression in patients is unknown.

The investigators' broad objective is to assess homocysteine metabolism and systemic endothelial function at the early stages of the disease and determine the prognostic value of homocysteine, related metabolites, and markers of endothelial function and injury to estimate renal disease severity and progression in patients with early ADPKD.

Participants in this study will have a blood and a urine sample collected to determine biomarkers of oxidative stress, endothelial function and injury, homocysteine, and related metabolite levels. In addition, peripheral arterial tonometry (PAT) will determine systemic endothelial function, and an abdominal MRI will be performed to determine the patient's total kidney volume (TKV).

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects, 15-40 years of age, inclusive
* Previous diagnosis of ADPKD (Based on Ravine et al. criteria)
* Class 1 according to imaging classification
* Estimated GFR>70 mL/min/1.73m^2(CKD-EPI)
* Ability to provide written, informed consent.

Exclusion Criteria:

* Class 2 according to imaging classification
* A concomitant systemic disease affecting the kidney
* Diabetes mellitus
* Predicted urine protein excretion in urinalysis >1 g/24 hrs
* Subjects having contraindications to or interference with MRI assessments
* Patients that are part of an interventional study or taking tolvaptan
* Female subjects that are pregnant

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female patients with a previous diagnosis of ADPKD that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in height adjusted Total kidney volume (htTKV) | Baseline to 24 months
  TKV determined by MRI
Baseline endothelial function, homocysteine and related metabolite levels as predictors of change in TKV | Baseline to 24 months
  Endothelial function determined by PAT and biochemical markers, TKV determined by MRI

SECONDARY OUTCOMES:
Change in systemic endothelial function | Baseline to 24 months
  Endothelial function determined by PAT
Change in biochemical markers related to endothelial function and injury | Baseline to 24 months
  Determined by ELISA and/or biochemical assays
Change in homocysteine and related metabolite levels | Baseline to 24 months
  Determined by 1HNMR, Mass spect, ELISA
Change in Renal blood flow (RBF) | Baseline to 24 months
  Determined by MRI
Change in estimated Glomerular filtration rate (GFR) | Baseline to 24 months
  eGFR determined by CKD-epi equation
NADPH oxidase 4 (NOX4) expression/activity | Baseline to 24 months
  Determined by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Maria V Irazabal, M.D.;Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study information — https://www.mayo.edu/research/clinical-trials/cls-20520136